CLINICAL TRIAL: NCT00693329
Title: Neutrophil Gelatinase-associated Lipcalin(NGAL): A Novel Blood Marker for Determining the Risk of Developing Contrast-Induced Nephopathy
Acronym: ENCINO
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Kyle Fortner, CRA, Biosite
Other Study IDs: BSTE-0406
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Cardiovascular Surgery With Coronary Angiography
Keywords: Contrast Induced Nephrophathy (CIN); Kidney; NGAL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample taken at 8 timepoints over 2 days.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a multi-center clinical study designed to assess the performance of the Triage NGAL test as an aid in the early risk assessment for contrast-induced nephropathy (CIN). Approximately 260 adults at risk for CIN undergoing intra-arterial angiography involving administration of iodinated contrast agent(s) will be enrolled.

DETAILED DESCRIPTION:
EDTA anti-coagulated blood samples will be drawn at eight different time points from within 1 hour prior to first contrast administration through 48 hours. These blood samples will be processed to plasma at the clinical site, frozen and shipped to Biosite for storage and testing of Triage NGAL and serum creatinine. The results of these assessments will be blinded to the medical team during the study and will not impact the medical management of the subject.

Any additional serum creatinine measurements obtained by the medical team as part of routine care as well as need for dialysis, hospitalization, major adverse cardiovascular events and mortality will be recorded through Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older;
* Undergoing angiographic procedure involving the intra-arterial administration of iodinated contrast agent(s);
* Chronic kidney disease indiacated by an eGFR < 75 ml/min/1.73 m2 based on screening labs performed ≤ 3 months prior to procedure.
* Able and willing to provide written informed consent for study participation and to comply with all study procedures.

Exclusion Criteria:

* Renal transplant recipients
* Pre-existing evidence of acute renal failure at the time of enrollment.
* Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at enrollment.
* Coronary artery bypass surgery or PCI within the previous 30 days.
* Participation in an interventional clinical study with an experimental therapy within the previous 30 days.
* Administration of intravasular contrast within the previous 30 days.
* Undergoing renal artery stenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing intra-arterial angiography involving administration of iodinated contrast agent(s).
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter McCullough, MD, Principal Investigator — Corewell Health East
Locations (3):
- United States (3):
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Providence Hospital, Providence, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan